CLINICAL TRIAL: NCT02685280
Title: Feasibility Study Regarding the Implantation and Use of Rechargeable Neurostimulators in Deep Brain Stimulation for Psychiatric Disorders (Either Obsessive-compulsive Disorder or Major Depression)
Brief Title: Rechargeable Neurostimulators in Deep Brain Stimulation for Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S50760; B32220072682 (Other: Belgian national government)
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Obsessive-compulsive Disorder; Depression
Keywords: rechargeable neurostimulators
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DBS for psychiatric disorders patients (Experimental): Patients on deep brain stimulation for either obsessive-compulsive disorder or major depression, undergoing rechargeable neurostimulator implantation as intervention
  Interventions: Device: Medtronic Restore Advanced 37713

INTERVENTIONS:
Device: Medtronic Restore Advanced 37713 — Rechargeable neurostimulators are implanted when the non-rechargeable neurostimulators are end-of-life.
  Other Names: Medtronic Restore 37711; Medtronic Activa RC 37612

SUMMARY:
From 1999 onwards, Deep Brain Stimulation [DBS] has been proposed as an alternative to capsulotomy in refractory cases of Obsessive-Compulsive Disorder [OCD]. More recently, several studies with DBS in patients with major depression have been initiated. In Belgium, there is currently a reimbursement for devices for DBS for OCD, but not for rechargeable neurostimulators, in these OCD patients.

Although rechargeable neurostimulators are widely used in spinal cord stimulation for pain and DBS for movement disorders, they have not yet been used in DBS for psychiatric disorders population. Several possible problems might arise with the use of rechargeable neurostimulators in this highly specific population.

In this prospective study with a before-after design, we would like to determine if the use of rechargeable neurostimulators is effective, applicable and safe and capable of diminishing the need for neurostimulator replacement procedures.

DETAILED DESCRIPTION:
BACKGROUND

Obsessive-Compulsive Disorder [OCD] is a psychiatric disorder with a lifetime prevalence of 2% which is mainly characterized by obsessional ideas and compulsive behaviours and rituals. Many patients show improvement under cognitive behavioural and/or pharmacological treatment. A minority of patients is refractory to all available therapy and may benefit from capsulotomy1.

From 1999 onwards, Deep Brain Stimulation [DBS] has been proposed as an alternative to capsulotomy in refractory cases of OCD (2,3). In Belgium, there is currently a reimbursement for devices for DBS for OCD, but not for rechargeable neurostimulators, in these OCD patients.

STUDY RATIONALE

Some patients with DBS for OCD need very frequent replacements of their neurostimulators (Medtronic Synergy 7427 ® [Synergy], Medtronic Kinetra 7428 ® [Kinetra] , Medtronic Activa PC 37601 ® [Activa PC] ), due to end-of-life of the batteries. This results in frequent re-interventions, probably causing discomfort for the patient, wound problems and infections due to revision surgery scar tissue, hardware problems and increasing costs for the public health system (consultations, hardware devices, surgery and its complications).

A new type of neurostimulators with an externally rechargeable battery has been developed recently. The manufacturer estimates the longevity of these devices to be 9 years. These products are in conformity with the essential requirements of Directive 1999/5/EC on Radio and Telecommunications Terminal Equipment and Directive 90/385/EEC on Active Implantable Medical Devices. Currently they have a CE mark only for the indication of DBS for Parkinson's Disease and Essential Tremor, but not for DBS for psychiatric disorders such as OCD. Therefore, up till now they cannot be used in patients treated with DBS for OCD.

Therefore, this physician-initiated study is trying to investigate whether the use of this new rechargeable neurostimulator is effective and safe in DBS treated OCD patients.

HYPOTHESIS

The hypothesis of the present study is that the implantation and use of rechargeable neurostimulators in OCD patients treated with DBS is (1) effective, (2) applicable, (3) safe and (4) decreases the need of neurostimulator replacement.

OBJECTIVES

To prove the hypothesis, the following objectives are aimed in our study:

1. Efficacy:

   -To test whether DBS using rechargeable neurostimulators is effective on psychiatric symptoms as compared to DBS using non-rechargeable neurostimulators in these patients.
2. Applicability:

   -To investigate whether this specific patient population is capable of recharging the rechargeable neurostimulators properly.
3. Safety:

   -To document possible side effects of DBS for OCD using rechargeable neurostimulators.
4. Capability of diminishing the need of neurostimulator replacement:

   -To investigate whether discomfort and risks of the frequent neurostimulator replacements due to battery end-of-life can be diminished by the use of the rechargeable neurostimulators.

   STUDY DESIGN

   At the Neurosurgery and Psychiatry consultation, eligible patients are informed about the present study. As soon as informed consent is obtained, the next time the battery of the non-rechargeable neurostimulator reaches its end-of-life and elective replacement is planned, a rechargeable neurostimulator and (if needed) the extension leads adaptors necessary to connect these neurostimulators with the existing extension leads will be implanted instead of a new non-rechargeable neurostimulator.

   After informed consent is obtained, at every consultation before and after implantation of the rechargeable neurostimulator the parameters as stated in the primary and secondary endpoints' sections will be recorded.

   TRIAL INTERVENTION

   The main trial intervention of this study will be the implantation of one rechargeable neurostimulator instead of the currently used non-rechargeable neurostimulator(s) and surgical closure of one of the existing abdominal wall cavities (the so-called "pockets"). It may be necessary to tunnel the extension cable from one side to another within the thoracic or abdominal wall. Thereby, we may provoke extension cable loops which may provoke undesirable stimulation when passing through a magnetic field. However this risk seems smaller than the risk of dissecting the electrode and replacing the extension cable to the other side.

   This intervention can be done under general or local anaesthetics.

   ADVERSE EVENTS REPORTING

   All adverse events are noted before and after implantation of the rechargeable neurostimulator.

   Below is a list of possible adverse events with both non-rechargeable and rechargeable neurostimulators for DBS in OCD:
   * Early and late surgery and anaesthesia related problems

     * A "pulling" experience at the level of the implanted neurostimulator and extension cables
     * Postoperative pain and discomfort
     * Displacement of the neurostimulator
     * Erosion of the skin superficial to the implanted hardware
     * Allergic reaction or rejection towards the implanted hardware
     * Wound infection and infection of the implanted hardware
     * Swelling or hematoma in the region of implantation
     * Pain, itching or discomfort at incision/implant sites
     * Death
   * Hardware and directly stimulation-related problems

     * Hardware failure (e.g. breakage or isolation damage of a cable, neurostimulator failure…)
     * Unwanted spontaneous reset of the neurostimulator
     * Fluctuating results
     * Early end-of-life (less than expected) of the battery of the neurostimulator
     * Playing with patient programmer
     * Shocking or jolting stimulation
     * Exceeding of the upper limit of current that is passed through the DBS system, as indicated by the manufacturer, that in extreme circumstances might lead to a biological effect at the tip of the electrode that is comparable to capsulotomy
     * Electromagnetic interference might lead to dysfunction of the DBS system and in extreme circumstances even to death (e.g. during MRI scanning)
   * Motor and movement problems

     * Teeth grinding
     * Akathisia
     * Balance disturbance
     * Coordination problems
     * Torticollis
     * Cheek twitches
     * Other muscle contractions
     * Increased tics
     * Fractures
     * Tremor
   * Sleeping problems and fatigue

     * Insomnia
     * Hypersomnia
     * Increased fatigue
     * Vivid dreams and nightmares
   * Gastro-intestinal problems

     * Altered sensation of taste/smell
     * Weight gain or weight loss
     * Nausea and vomiting
     * Increased hungriness or decreased appetite
     * Esophagitis
     * Slow gastric emptying
     * Abdominal pain
     * Diarrhoea or constipation
     * Anal blood loss
   * Mouth, ENT and respiratory problems

     * Nose bleed
     * Dental infections
     * Dry mouth
     * Tinnitus
     * Hump of earwax
     * Respiratory infection
     * Shortness of breath
     * Sleep apnoea
   * Sexual and urinary problems

     * Urinary, prostate or kidney infection
     * Libido increase or decrease
     * Erection decrease
     * Ejaculation problem
     * Vaginal discharge
     * Urinary incontinence
     * Increased urinary frequency
   * Cardiovascular problems

     * Palpitations
     * Arterial hypertension
     * Episodic retrosternal pain
   * Neurologic problems

     * Headaches
     * A "flashing" sensation in the head
     * Pain away from incision/implant sites
     * Dizziness
     * Sedation
     * Paraesthesia
     * Changes in handwriting
     * Perseveration
     * Seizures
     * Coma
     * Paralysis
   * General problems

     * Transpiration
     * Warm and cold feeling
     * Nail biting
     * Body smell change
     * Hair pulling
     * Hair loss
     * Skin and skin attachment infection
   * Laboratory test abnormalities

     * Increased creatine kinase
     * Low ferritine
     * Increased amylase
     * Hypercholesterolemia
     * Diabetes mellitus
   * Psychiatric and cognitive problems

     * Irritability
     * Suicidality (thoughts/attempts)
     * Increased depression
     * Increased anxiety
     * Increased OCD
     * Aggression/violent behaviour
     * Angry
     * Overdrive
     * Memory complaints
     * Disinhibition
     * Recklessness
     * Hyperactivity
     * Logorrhoea
     * Accident proneness
     * Hypomania
     * Cognitive disturbance (clouding)
     * Panic attack
     * Tension/nervousness
     * Hysteria
     * Apathy
     * Loss of motivation
     * Lack of energy
     * Flashbacks
     * Confusion
     * Blackouts
     * Derealisation/depersonalisation
     * Excessive alcohol drinking
     * Medication abuse
     * Paranoia
     * Delusion
     * Family problems

   Below is a list of possible adverse events with rechargeable but not with nonrechargeable neurostimulators for DBS in OCD:
   * A heating sensation over the neurostimulator during recharging
   * Local skin irritation over the neurostimulator during or after recharging
   * Hardware failure of the recharger including breakage of the recharger fixation belt.
   * Insufficient quality of the connection for energy transfer between the rechargeable neurostimulator and the recharger.
   * The battery of the rechargeable stimulator always needs to be recharged before it is totally empty. After more than one episode of a totally empty battery further proper functioning of the neurostimulator nor replacement within the proposed study design cannot be guaranteed by the constructor.

   A committee consisting of the principle investigators will decide whether an adverse event is definitely, probably, possibly or not an adverse event due to the system for DBS for OCD. All expected and unexpected adverse events will be noted and published.

   BIOSTATISTICS AND DATA ANALYSIS

   Paired statistical tests for continuous data (A, f, PW, number of consultations,) and for ordinal data (Y-BOCS, GAF, HAM-A, HAM-D, BDI) pre- and post-implantation, as well as descriptive statistics for continuous data (number of recharging sessions, number of battery status controls, battery longevity, preferred stimulator type at replacement), will be used. No power calculation is performed.

   ETHICS

   Approval of the UZ/KU Leuven Ethics Committee, working after the ICH-GCP principles, will be asked for. All data will be collected in an objective, careful and precise manner.

   All risks will be kept as low as possible with a meticulous implantation procedure and a careful clinical evaluation before and after implantation. Participation in the study is completely voluntary.

ELIGIBILITY:
Inclusion Criteria:

* DBS for OCD / DBS for MD patients, AND
* experiencing a beneficial effect of DBS on the psychiatric symptoms, AND
* needing at least 1 IPG replacement per 18 months, AND
* in the possibility to give informed consent for this study

Exclusion Criteria:

* anyone not meeting all the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Y-BOCS (for OCD) | from 2 years before intervention until 2 years after intervention
  Change in mean Yale-Brown Obsessive Compulsive Scale (Y-BOCS). Mean Y-BOCS during the first 2 years after intervention minus mean Y-BOCS during the last 2 years before intervention.
Change in HAM-D (for MD) | from 2 years before intervention until 2 years after intervention
  Change in Hamilton Depression Rating Scale (HAM-D). Mean HAM-D during the first 2 years after intervention minus mean HAM-D during the last 2 years before intervention.

SECONDARY OUTCOMES:
Change in HAM-D (for OCD) | from 2 years before intervention until 2 years after intervention
  Change in Hamilton Depression Rating Scale (HAM-D). Mean HAM-D during the first 2 years after intervention minus mean HAM-D during the last 2 years before intervention.
Change in BDI | from 2 years before intervention until 2 years after intervention
  Change in Beck Depression Inventory (BDI). Mean BDI during the first 2 years after intervention minus mean BDI during the last 2 years before intervention.
Change in GAF | from 2 years before intervention until 2 years after intervention
  Change in Global Assessment of Functioning (GAF). Mean GAF during the first 2 years after intervention minus mean GAF during the last 2 years before intervention.
Change in Stimulation Amplitude | from 2 years before intervention until 2 years after intervention
  Change in Stimulation amplitude as measured in volt. Mean stimulation amplitude during the first 2 years after intervention minus mean stimulation amplitude during the last 2 years before intervention.
Change in Stimulation Frequency | from 2 years before intervention until 2 years after intervention
  Change in Stimulation frequency as measured in hertz Mean stimulation frequency during the first 2 years after intervention minus mean stimulation frequency during the last 2 years before intervention
Change in Pulse Width | from 2 years before intervention until 2 years after intervention
  Stimulation pulse width as measured in seconds. Mean stimulation pulse width during the first 2 years after intervention minus mean stimulation pulse width during the last 2 years before intervention.
Change in Contact Configuration | from 2 years before intervention until 2 years after intervention
  Change in stimulation contact configuration as expressed in fraction of patients using a certain contact point as anode or cathode.
  Fraction of patients using a certain contact point as cathode or anode during the first 2 years after intervention minus fraction of patients using a certain contact point as cathode or anode during the last 2 years before intervention.
Change in frequency of outpatient clinic contacts at the Psychiatry department | from 2 years before intervention until 2 years after intervention
  Change in frequency of outpatient clinic contacts at the Psychiatry department. Frequency of outpatient clinic contacts at the Psychiatry department during the first 2 years after intervention minus frequency of outpatient clinic contacts at the Psychiatry department during the last 2 years before intervention.
Change in fraction of hospitalized days at the Psychiatry department | from 2 years before intervention until 2 years after intervention
  Change in fraction of hospitalized days at the Psychiatry department. Fraction of hospitalized days at the Psychiatry department during the first 2 years after intervention minus fraction of hospitalized days at the Psychiatry department during the last 2 years before intervention.
Change in frequency of outpatient clinic contacts at the Neurosurgery department | from 2 years before intervention until 2 years after intervention
  Change in frequency of outpatient clinic contacts at the Neurosurgery department.
  Frequency of outpatient clinic contacts at the Neurosurgery department during the first 2 years after intervention minus frequency of outpatient clinic contacts at the Neurosurgery department during the last 2 years before intervention.
Change in fraction of hospitalized days at the Neurosurgery department | from 2 years before intervention until 2 years after intervention
  Change in fraction of hospitalized days at the Neurosurgery department. Fraction of hospitalized days at the Neurosurgery department during the first 2 years after intervention minus fraction of hospitalized days at the Neurosurgery department during the last 2 years before intervention.
Change in frequency of DBS-related surgical procedures | from initial electrode implantation through study completion (on average approximately 5 years)
  Change in frequency of neurosurgical procedures related to the DBS system. Frequency of neurosurgical procedures related to the DBS system after intervention minus frequency of neurosurgical procedures related to the DBS system before intervention.
Adverse events | from initial electrode implantation through study completion (on average approximately 5 years)
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bart Nuttin, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No